CLINICAL TRIAL: NCT06799572
Title: The Effect of Massage on Pain, Comfort and Feeding Status of Preterm Infants Under Nasal Continuous Positive Airway Pressure (NCPAP)
Brief Title: The Effect of Massage on Preterm Babies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem BOZBUĞA (Other)
Responsible Party: Sponsor-Investigator, Özlem BOZBUĞA, Msc. Nurse, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OBOZBUGA-1
Record Dates: First submitted 2025-01-11; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: PreTerm Neonate; nCPAP; Massage
Keywords: ncpap; massage; preterm
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Intervention Model Description: This research will be carried out as a randomised controlled experimental study in a pretest-posttest design in order to examine the effect of massage on pain, comfort and nutritional status of preterm infants who received Ncpap in the neonatal intensive care unit. ClinicalTrials number will be obtained for the research.Preterm infants will be randomly assigned to the study groups according to gestational week at birth and gender using a computer programme (randomizer.org). Power analysis was used to calculate the sample size of the randomised controlled trial. G*Power 3.1.9.7. programme with 95% power, 0.05 error margin and 2.23 effect size, the sample size was calculated as 12 people for each group. Considering the loss of data in the study, it was decided to include 15 people in each group. The reference study was used to determine the effect size [16]Preterm infants in the experimental and control groups will be selected similarly according to sex, birth weight, gestational week,
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- massage group (Experimental): * A follow-up form and scales will be applied to the babies before the first massage session.
  * Massage will be applied by the researcher in the incubator for 15 minutes
  * Massage will be done twice a day, morning and evening
  * Babies will be massaged for a total of 5 days (10 sessions)
  * In the massage to be applied to babies, liquid petroleum jelly will be used to provide lubrication on the skin. Vaseline is recommended for newborn skin care because it is the most effective, reliable and inexpensive. [19, 20].
  * After 10 sessions of massage, Pain and Comfort scales will be applied and the final evaluation of the follow-up form will be made.
  * Each massage will be performed 1 hour after feeding.
  * Data such as vomiting, distension, defecation frequency, etc. of the baby the day before will be recorded on the Newborn Monitoring Form before the morning massage to be performed every day.
  * NIPS pain assessments of preterm babies will be performed after the procedure
  Interventions: Other: massage
- control group (No Intervention): Follow-up form, pain and comfort scales will be applied simultaneously with the experimental group.

INTERVENTIONS:
Other: massage — Hands will be washed with hand soap and rubbed with disinfectant before the procedure.
  * The head of the bed is raised by 30°-45° in the incubator.
  * The baby is placed face down.
  * Vaseline is applied to the hands.
  * The 15 minute session will consist of three 5 minute phases. Phase 1 will be tactile stimulation phase, Phase 2 will be kinesthetic stimulation and Phase 3 will be I Love You technique.
  * In the tactile stimulation phase, the infant is turned to the prone position and a stroking motion (12 strokes in approximately 5 seconds) will be applied with moderate pressure in 1-minute intervals, from the top of the head to the neck and back to the top of the head, from the neck to the shoulder, from the neck to the shoulder, from the upper back to the waist and back to the upper back, from the thigh to the foot and both legs, from the shoulder to the hand and from both arms to the shoulder.
  * In the kinesthetic stimulation phase, the infant is placed in the supine position and eac
  Arms: massage group

SUMMARY:
This study was planned as a randomized controlled experimental study with pre-test post-test design in order to examine the effect of massage on pain, comfort and nutritional status in infants undergoing NCPAP in the NICU, considering that massage may be effective in reducing the effectiveness of treatment and complications that may develop due to NCPAP by reducing stress in newborns undergoing NCPAP.In this research, answers to the following questions will be sought; Massage has an effect on pain in preterm infants receiving NCPAP therapy; H1: has an effect on pain. H2: has an effect on comfort. H3: has an effect on feeding intolerance (vomiting, abdominal distension, stool output...)

DETAILED DESCRIPTION:
1. Introduction Neonatal intensive care unit (NICU) is a place where postnatal babies are followed up due to respiratory distress, sepsis, congenital anomalies, prematurity and the problems caused by it. With the advances in technology and science, the survival rate of preterm babies has increased, but morbidity is increasing. Respiratory failure, which is associated with high neonatal morbidity and mortality, is a common clinical condition that negatively affects newborns according to their gestational age. Respiratory distress is generally seen physiologically due to the immaturity of the lungs of preterm infants and mechanical ventilation application support is needed. Nasal continuous positive airway pressure (NCPAP), which is most commonly used as initial treatment, is a treatment method used to provide respiratory support in preterm infants. NCPAP increases the pressure in the lungs by providing preterm babies with a continuous airflow through the nasal passage (with mask / cannula), prevents airway closure, prevents air trapping in the lungs and supports breathing. However, undesirable conditions such as pain, gastric distension, feeding intolerance, nasal injury and pneumothorax may occur in preterm infants with NCPAP application. Nonpharmacological methods such as positioning and massage can be used to prevent these complications, to increase the comfort of infants during treatment and to obtain a positive response to treatment. Massage reduces stress and pain, increases vagal activity, gastric motility and weight gain in newborns increases the frequency of defecation reduces the level of bilirubin has been reported. It has been determined that massage decreases stress levels in newborns monitored on mechanical ventilator, regulates respiratory rhythm with relaxant effect and increases the effectiveness of treatment.

   When the literature was examined, although there were studies evaluating the effectiveness of massage in the neonatal unit . The study evaluating the effect of massage in preterm infants receiving NCPAP is limited. This study was planned as a randomised controlled experimental study with pre-test post-test design in order to investigate the effect of massage on pain, comfort and nutritional status in infants undergoing NCPAP in the NICU, considering that massage may be effective in reducing the effectiveness of treatment and complications that may develop due to NCPAP by reducing stress in newborns undergoing NCPAP.
2. MATERIALS AND METHODS 2.1.Purpose and Type of Research This research will be carried out as a randomised controlled experimental study in a pretest-posttest design in order to examine the effect of massage on pain, comfort and nutritional status of preterm infants who received Ncpap in the neonatal intensive care unit.

2.2. Hypotheses of the Research Massage in preterm infants receiving NCPAP therapy; H1 : has an effect on pain. H2 : has an effect on comfort. H3 : has an effect on nutritional intolerance (vomiting, abdominal distension, faecal output...).

2.3. Variables of the Research The independent variables of the study were the variables included in the Form of Descriptive Characteristics of Newborns (birth weight, gestation week and sex of the baby...).

The dependent variables of the study were pain and comfort scale scores of preterm infants, feeding intolerance status (presence of vomiting, abdominal distension, number of stools/day).

2.4. Location of the Research The study will be conducted in the NICU of Health Sciences University Adana City Training and Research Hospital. There are 4 neonatologists, 6 assistant doctors and 69 nurses working in the NICU.

2.5. Population and Sample of the Study The population of the study will consist of infants who underwent NCPAP due to respiratory distress in the NICU of Adana City Training and Research Hospital. Preterm infants will be randomly assigned to the study groups according to gestational week at birth and gender using a computer programme (randomizer.org). Power analysis was used to calculate the sample size of the randomised controlled trial. G*Power 3.1.9.7. programme with 95% power, 0.05 error margin and 2.23 effect size, the sample size was calculated as 12 people for each group. Considering the loss of data in the study, it was decided to include 15 people in each group. The reference study was used to determine the effect size. All stages of randomised controlled trials should be conducted according to the Consolidated Standards of Reporting Trials (CONSORT).

Inclusion Criteria; Infants of parents who agreed to participate in the study,

* Receiving NCPAP therapy for at least 1 day,
* Gestational age greater than 32 weeks
* Birth weight over 1500 grams
* Infants fed with orogastric + total parenteral nutrition (TPN) will be included.

Exclusion Criteria;

* Infants with necrotising entecolitis, suspected or confirmed sepsis,
* No skin disease,
* Not receiving sedation (considering that it may affect pain response),
* Babies who have undergone surgical intervention (abdominal and central nervous system, cardiac surgery)
* Babies of substance-abusing mothers,
* Infants of parents who do not agree to participate in the study will not be included.

Exclusion criteria; Babies in the massage group who switched from Ncpap to IMV, who underwent surgical intervention with sedation and who developed NEC will be excluded from the study.

Criteria for Matching Working Groups Preterm infants in the experimental and control groups will be selected similarly according to sex, birth weight, gestational week, postnatal age and mode of delivery.

2.6. Data Collection Tools 2.6.1. Newborns' Descriptive Characteristics Form (Annex 3) This form includes information such as gestation week, sex, birth weight, postnatal day, etc. of newborns.

2.6.2. Newborn Monitoring Schedule (Annex 4) This form is a daily monitoring form in which the baby's daily weight gain, feeding pattern, vomiting and abdominal distension, and the number of stools will be recorded.

2.6.3. Neonatal Pain Scale (Appendix -5) Neonatal Infant Pain Scale (NIPS) was developed by Lawrence et al. (1993). It was adapted into Turkish by Akdovan (1999). It is a pain assessment scale developed for premature and newborns and behaviourally evaluates the response to pain in invasive procedures. The total score in NIPS varies between 0 and 7, and scores higher than 3 indicate the presence of pain. (Akdovan, 1999). Six behavioural categories are assessed, with a minimum score of 0 and a maximum score of 7. High validity and reliability (r= .84-.92) (17) 2.6.4.Newborn Comfort Behaviour Scale (Appendix-6) The Turkish validity and reliability study of the Neonatal Comfort Behaviour Scale (NCCS) was conducted by Kahraman et al. in 2014. The NBBS is a Likert-type scale consisting of 6 parameters including alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. In newborns receiving mechanical ventilator support, the item "Respiratory Response" is evaluated and in those not receiving mechanical ventilator support, the item "Crying" is evaluated. In the validity and reliability study of the scale, Cronbach's alpha coefficient was found to be 0.85 for the primary researcher and 0.82 for the assistant researcher before care and 0.92 for the primary researcher and 0.85 for the assistant researcher after care. The score that can be obtained from the scale is between 6-30. If the total score of the scale is between 9-13, the baby is comfortable; if it is between 14-30, it shows that the baby has pain or distress, the baby is uncomfortable and needs interventions to provide comfort.

2.8. Implementation of the Research The families of the infants who meet the inclusion criteria will be informed about the purpose, content and method of the study, and verbal and written consent (Appendix 8, 9: Informed Voluntary Consent Form) will be obtained from the parents who agree to participate in the study. Descriptive characteristics form, patient follow-up form and scales will be completed before the procedure for the babies in both groups.

Experimental group: In this study, preterm infants who were included in the massage group will be massaged twice a day (morning and evening) for 5 days, each session lasting 15 minutes. The babies included in the study will be monitored by the researcher for 5 days in the morning and evening as follows. Weighing in the clinic is done in the evening.

Experimental group:

* A follow-up form and scales will be applied to the babies before the first massage session.
* Massage will be applied by the researcher in the incubator for 15 minutes
* Massage will be done twice a day, morning and evening
* Babies will be massaged for a total of 5 days (10 sessions)
* In the massage to be applied to babies, liquid petroleum jelly will be used to provide lubrication on the skin. Vaseline is recommended for newborn skin care because it is the most effective, reliable and inexpensive.
* After 10 sessions of massage, Pain and Comfort scales will be applied and the final evaluation of the follow-up form will be made.
* Each massage will be performed 1 hour after feeding.
* Data such as vomiting, distension, defecation frequency, etc. of the baby the day before will be recorded on the Newborn Monitoring Form before the morning massage to be performed every day.
* NIPS pain assessments of preterm babies will be performed after the procedure.

Control group:

- Follow-up form, pain and comfort scales will be applied simultaneously with the experimental group.

2.9. Evaluation of Data In the evaluation of the data obtained from the study, statistical package programme (IBM SPSS 24.0) will be used in computer environment and significance will be evaluated at p<0.05 level.

2.10. Ethical Dimension of the Research Ethics committee permission was obtained from Health Sciences University Adana City Hospital Ethics Committee and institutional permission (30.05.2024/17-1) was obtained from Adana City Hospital. Consent will be obtained from the parents of the babies to be included in the study. In addition, permission was obtained via e-mail for the use of the scales to be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Infants of parents who agreed to participate in the study,

  * Receiving NCPAP therapy for at least 1 day,
  * Gestational age greater than 32 weeks
  * Birth weight over 1500 grams
  * Infants fed with orogastric + total parenteral nutrition (TPN) will be included.

Exclusion Criteria:

* • Infants with necrotising entecolitis, suspected or confirmed sepsis,

  * No skin disease,
  * Not receiving sedation (considering that it may affect pain response),
  * Babies who have undergone surgical intervention (abdominal and central nervous system, cardiac surgery)
  * Babies of substance-abusing mothers,
  * Infants of parents who do not agree to participate in the study will not be included.

Babies in the massage group who switched from Ncpap to IMV, who underwent surgical intervention with sedation and who developed NEC will be excluded from the study.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | 5 day
  Neonatal Infant Pain Scale (NIPS) was developed by Lawrence et al. (1993). It was adapted into Turkish by Akdovan (1999). It is a pain assessment scale developed for premature and newborns and behaviourally evaluates the response to pain in invasive procedures. The total score in NIPS varies between 0 and 7, and scores higher than 3 indicate the presence of pain. (Akdovan, 1999). Six behavioural categories are assessed, with a minimum score of 0 and a maximum score of 7. High validity and reliability (r= .84-.92)
Daily Monıtoring Form | 5 day
  This form is a daily monitoring form in which the baby's daily weight gain, feeding pattern, vomiting and abdominal distension, and the number of stools will be recorded
Neonatal Comfort Behaviour Scale (NCCS) | 5 day
  The Turkish validity and reliability study of the Neonatal Comfort Behaviour Scale (NCCS) was conducted by Kahraman et al. in 2014. The NBBS is a Likert-type scale consisting of 6 parameters including alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. In newborns receiving mechanical ventilator support, the item "Respiratory Response" is evaluated and in those not receiving mechanical ventilator support, the item "Crying" is evaluated. In the validity and reliability study of the scale, Cronbach's alpha coefficient was found to be 0.85 for the primary researcher and 0.82 for the assistant researcher before care and 0.92 for the primary researcher and 0.85 for the assistant researcher after care. [18]. The score that can be obtained from the scale is between 6-30. If the total score of the scale is between 9-13, the baby is comfortable; if it is between 14-30, it shows that the baby has pain or distress, the baby is uncomfortab

CONTACTS AND LOCATIONS:
Overall Officials: EMİNE ERDEM, Study Chair — TC Erciyes University; OZNUR BASDAS, Study Director — TC Erciyes University; SELVİ GULAŞI, Study Director — Adana City Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No